CLINICAL TRIAL: NCT05485038
Title: General Anesthesia Versus Awake Surgery in Resection of Gliomas and Metastases of Motor Areas: a Randomised, Controlled Trial
Brief Title: General Anesthesia Versus Awake Surgery in Resection of Gliomas and Metastases of Motor Areas
Acronym: GAMMA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Principal Investigator, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9d
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gliomas Benign; Glioma, Malignant; Metastases to Brain
Keywords: contrast-enhancing glioma; non-enhancing glioma; brain metastasis; awake surgery; general anesthesia; motor area
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Dynamics of motor function before, within 10 days after surgery and in 3 months after surgery will be assessed by neurosurgeon blinded for the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Awake surgery (Experimental): Critical steps of brain mapping and tumor removal will be performed in awake patient
  Interventions: Procedure: Tumor resection in awake patient
- General anesthesia (Active Comparator): Brain mapping and tumor removal will be performed in asleep patient
  Interventions: Procedure: Tumor resection in asleep patient

INTERVENTIONS:
Procedure: Tumor resection in awake patient — Surgeon performs critical steps of tumor removal in awake patient and controls his/her motor functions by brain mapping and assessing of voluntary movements
  Arms: Awake surgery
Procedure: Tumor resection in asleep patient — Surgeon removes tumor in asleep patient and controls his/her motor functions by brain mapping
  Arms: General anesthesia

SUMMARY:
Objective of the study is to determine whether resection of gliomas and metastases of motor areas using awake surgery can achieve rarer motor deterioration after operation than using general anesthesia.

DETAILED DESCRIPTION:
Awake surgery is usually used for tumor resection located in language areas. But patient's awakening during removal of mass lesions from motor areas can give additional opportunities. Besides checking of muscle contractions and integrity of motor fibers a surgeon in awake patient can assess planning of movements, praxis, visual feedback and vestibular processing of motions. Preserving of voluntary movements can be an additional proof that cortical motor centers and corticospinal tract were not damaged. At the moment there are no published results of randomized trials showing advantage of awake surgery in removal of mass lesions from motor brain areas.

Objective of the study is to determine whether resection of gliomas and metastases of motor areas using awake surgery can achieve rarer motor deterioration after operation than using general anesthesia.

Participants of the study will be randomly operated using awake surgery or general anesthesia. In both groups intraoperative neuromonitoring will be used. Dynamics of motor functions will be assessed before and after surgery by blinded neurologists.

ELIGIBILITY:
Inclusion Criteria:

* single gliomas without contrast enhancement in preoperative magnetic resonance imaging (presumed low-grade gliomas)
* single gliomas with contrast enhancement in preoperative magnetic resonance imaging (presumed high-grade gliomas)
* one or several brain metastases from any cancer
* location near primary motor area or corticospinal tract
* newly diagnosed
* Karnofsky Performance Status 60-100%
* muscle strength in assessed limbs 3-5 points in Medical Research Council scale
* age 18-69 years
* body mass index 29 and less
* hemoglobin 110 and more
* platelets 100 and more
* international normalized ratio less than 2,0
* presumed blood loss no more than 8-10 percents of circulating blood volume (no more than 450-650 milliliters)

Exclusion Criteria:

* chronic obstructive pulmonary disease
* persistent smoker (smoking index 11 and more)
* major comorbidities
* implanted pacemaker
* inability to perform intraoperative tests before surgery
* severe aphasia
* psychiatric disorders
* barely controlled seizures
* contraindications to magnetic resonance imaging
* previously performed brain radiotherapy
* pregnancy
* breast feeding

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite event of deterioration of early motor function, severe disturbance of consciousness or death from any cause | within 10 days after surgery
  Motor function is assessed in Medical Research Council scale and is compared before and after surgery, deterioration of motor function means decline of 1 grade or more; level of consciousness is assessed in Glasgow Coma scale, it's severe disturbance means decline to 9 points or less
Dynamics of early motor function (in grades) | within 10 days after surgery
  Early motor function is assessed in Medical Research Council scale and is compared before and after surgery
Dynamics of late motor function (in grades) | in 3 months after surgery
  Late motor function is assessed in Medical Research Council scale and is compared before and in 3 months after surgery

SECONDARY OUTCOMES:
Composite event of deterioration of early speech, severe disturbance of consciousness or death from any cause | within 10 days after surgery
  Speech function is assessed in Hendrix scale (2017) and is compared before and after surgery, deterioration of speech function means decline of 1 grade or more; level of consciousness is assessed in Glasgow Coma scale, it's severe depressing means decline to 9 points or less
Early speech function (in grades) | within 10 days after surgery
  Early speech function is assessed in Hendrix scale (2017)
Early Karnofsky performance status (in percents) | within 10 days after surgery
  Assesses patients' possibilities to self-service in Karnofsky Performance Status scale
Extent of resection (in percents) | within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100
Gross total resection (Yes or No) | within 48 hours after surgery
  Absence of tumor tissue in postoperative magnetic resonance imaging
Duration of surgery (in minutes) | Intraoperatively
  Duration of surgery from skin incision till last skin suture
Intraoperative blood loss (in milliliters) | Intraoperatively
  Blood loss from skin incision till last skin suture
Duration of stay in intensive care unit (in days) | From admission to intensive care unit after surgery till transfer to neurosurgical unit, up to 365 days
  How long patient was treated in intensive care unit
Duration of hospital stay (in days) | From admission to the hospital till hospital discharge, up to 365 days
  How long patient was treated in the hospital from admission till discharge
Cerebral complications | within 3 months after surgery
  Which cerebral complications arose after surgery
Somatic complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which somatic disorders arose after surgery
Repeated hospital admission (Yes or No) | within 3 months after surgery
  Whether repeated hospital admissions were required due to postoperative complications
Late speech function (in grades) | in 3 months after surgery
  Late speech function is assessed in Hendrix scale (2017)
Late Karnofsky performance status (in percents) | in 3 months after surgery
  Assessment of patients' possibilities to self-service in Karnofsky Performance Status scale

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No